CLINICAL TRIAL: NCT04533412
Title: Comprehensive Home-based Self-management Support for COPD Patients
Brief Title: Comprehensive Self-management Support for COPD Patients
Acronym: SAMBA COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: City Health Works (Other); Northwestern University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alex D Federman, Director of Research, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GCO 17-2407; R34HL143747 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: COPD; Self-management Behaviors
Keywords: chronic obstructive pulmonary disease; pulmonary rehabilitation; intervention; home-based; randomized controlled trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: For the intervention, community health workers will assess barriers to good self-management behaviors that lie within 4 domains: 1) social context, 2) physical health and functioning, 3) cognitive factors, and 4) psychological factors. They will work with participants for 6 months to help them work through their barriers to self-management of COPD. Participants can also participate in home-based pulmonary rehabilitation and can receive emergency pack/action pack medication for COPD exacerbations.
  The attention control is designed to isolate the impact of screening for self-management barriers. The attention control will consist of 4 visits by a COPD educator who will review a COPD education booklet.
  Participants are randomized based on COPD Assessment Test (CAT) scores: CAT <10 vs CAT >10
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research coordinators (RCs) and investigators are blinded to study randomization and treatment arm for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted self-management barrier support (Experimental): Intervention group - Targeted self-management barrier support, home-based pulmonary rehabilitation, and emergency medication with community health workers
  Interventions: Behavioral: Self-management barrier support
- Guided COPD education (Active Comparator): Control group - Guided COPD education with a COPD educator
  Interventions: Behavioral: Basic COPD Education

INTERVENTIONS:
Behavioral: Self-management barrier support — For the intervention, community health workers will assess barriers to good self-management behaviors that lie within 4 domains: 1) social context, 2) physical health and functioning, 3) cognitive factors, and 4) psychological factors. They will work with participants for 6 months to help them work through their barriers to self-management of COPD. Participants can also participate in home-based pulmonary rehabilitation and can receive emergency pack/action pack medication for COPD exacerbations.
  Arms: Targeted self-management barrier support
Behavioral: Basic COPD Education — The attention control will consist of 4 visits by a COPD educator to the home to review the COPD education booklet. During the first visit, this COPD educator will review the COPD 1-2-3 booklet in its entirety with the patient. During visits 2 and 3, the COPD educator will make a visit to "check in" with the patient, ask how they are doing with their respiratory symptoms, and review any sections of the COPD 1-2-3 booklet the patient chooses. The COPD educator will recommend visits every 2 months but the patient and COPD educator may choose to modify the interval as needed. If the patient appears to be experiencing worsening respiratory symptoms during any visit, the COPD educator will notify the patient's physician.
  Arms: Guided COPD education

SUMMARY:
The study team will adapt and expand an effective model of asthma self-management support for patients with chronic obstructive pulmonary disease (COPD). In this new model, community health workers will comprehensively screen for and address barriers to effective COPD self-management, including maladaptive coping behaviors, and guide patients through home-based pulmonary rehabilitation. Feasibility of the new model will be assessed in preparation for a fully powered, multisite randomized trial.

DETAILED DESCRIPTION:
Phase II will focus on intervention implementation and evaluation (months 13-36).

The research team will randomize 58 COPD patients (29 per arm) to the SaMBA-COPD intervention or an attention control and follow them for 9 months to assess health and self-management behavior (SMB) outcomes.

Intervention:

Step 1: Outreach and Engagement. The project manager will notify the City Health Works (CHW) supervisor when an eligible and consented patient is randomized to receive care the intervention and will provide the patient's name and contact information. The CHW will call the patient within 7 days of consent to schedule a home visit. The CHW will encourage caregivers to join all meetings.

Step 2: Intake. The CHW will perform an intake interview that includes collection of basic information about the patient and their health and healthcare, including medications, intended to enable them to understand their health problems and provide them with chronic illness self-management support.

Step 3: Symptom assessment, medication adherence, and inhaler technique. The CHW will assess the patients' symptoms, adherence to medications, and check inhaler technique following a standardized protocol, and correct errors in inhaler use if identified.

Step 4: SMB barrier screening with the Screener. The CHWs will assess barriers to good SMB that lie within 4 domains: 1) social context, 2) physical health and functioning, 3) cognitive factors, and 4) psychological factors. To assess elements in each domain, the study team will use questions drawn from validated surveys used in the study team's research and in the SAMBA screening tool. Screening questions are a part of the study intervention, of which they consented to in the research consent. Examples of barriers follow:

1. Social context. Factors include adequacy of social support, financial and access concerns (costs, insurance, pharmacy convenience), language and literacy skills, coping with illness, alcohol and drug use, and use of culturally-rooted therapies like herbals and spiritual remedies.
2. Physical health and functioning. These include physical functioning and medication concerns (e.g., side effects, multiple medications).
3. Cognition. The CHW will screen for cognitive impairment with the validated Quick mild cognitive impairment screen (QMCI) because cognitive impairment may challenge their ability to perform SMB.
4. Psychology. Factors include depression and anxiety, and maladaptive beliefs about COPD and COPD medications.

Step 5: Addressing identified barriers. Each identified barrier links to a menu of actions for the patient and CHW to employ to resolve or work around it. Other actions may be identified by patient or CHW and pursued if desired. Wherever appropriate, the CHW will engage the patient's physicians and or a social worker to enact some of the action steps. Examples of barriers follow:

1. Social context barriers. Examples of actions include enrolling the patient in the New York State pharmaceutical assistance program to reduce drug costs or ask physicians to consider generic or formulary approved alternatives. If retrieving or renewing prescriptions is a problem, the CHW may pick up the medication or arrange delivery. The CHW can contact the physician to request a renewal if needed, and refer the patient to a social worker for assistance with home aid services, entitlements, insurance matters, and assistance when second hand smoke is a problem.
2. Physical health and functioning barriers. Examples include asking the physician to consider reducing medicines if the patient finds the regimen too burdensome, requesting occupational or physical therapy to address physical limitations, or engaging the social worker to arrange transportation.
3. Cognition barriers. The study team will specifically target memory but also use strategies to compensate based on type of impairment, including medication organization, slower-paced and explicit verbal instructions, use of tangible external aids, repetition and teach-back, use of plain language, and guided imagery to reduce cognitive load. Such strategies have been shown to improve SMB in low-literacy populations. The CHW may have more frequent encounters (in-person, phone) with memory impaired patients. Daily cell phone text reminders are another option that patients can select when memory problems impact regular medication use.
4. Psychological barriers. The CHW will notify the PCP if a participant voluntarily divulges any feelings of depression or anxiety. The PCP may evaluate and treat or refer to a mental health specialist.

COPD action plan and medication rescue pack. The study team will obtain consent from each patient's primary care provider to have a pharmacist counsel patients about rescue medications (oral steroids and antibiotics, "rescue pack") to be used in the event of an exacerbation of COPD. This consent will be obtained at the time of obtaining consent from the physician to recruit the patient for study participation. If the physician provides consent to recruit the patient but refuses consent to counsel the patient about the rescue pack, the patient will receive all intervention components with the exception of rescue pack counseling by a pharmacist.

For patients for whom the study team have consent from the PCP to provide counseling about the rescue pack, the CHW will suggest to the patient that they meet with the pharmacist. The meeting will be voluntary. For patients who agree, a referral will be made to the pharmacist and a visit scheduled, to take place in a clinical setting. The pharmacist will counsel the patient on the use of the rescue pack. If the patient agrees to receive a rescue pack, the pharmacist will place an order in the Epic electronic health record for the rescue pack medications, then pend and route the order to the patient's PCP. The PCP can choose to sign the order, cancel or delete it. The pharmacist will check to determine whether the prescription order was signed by the PCP. If it was not, the pharmacist will assume that the physician does not wish to provide the patient a rescue pack prescription. If the prescription order was signed by the physician, the pharmacist will contact the patient 7-10 days later to determine whether the patient picked up the medication and to ensure that the patient understands when and how to use the medications appropriately, and will notify the CHW that the patient received the medications. The CHW will discuss the use of the rescue pack medications with the patient at subsequent encounters to ensure that they continue to understand how to use them appropriately. Should the patient use the medications, the CHW, pharmacist, and or patient will notify the PCP, who will be encouraged to follow up with the patient.

Step 6: Home-Based Pulmonary Rehabilitation Protocol (HBPR). HBPR will be available to all patients who are able to ambulate with or without an assistive device (cane or walker), regardless of supplemental oxygen use. If the patient expresses interest in HBPR, the CHW will schedule the appointment and accompany the patient and caregiver (if available) to a clinical practice at the Mount Sinai Hospital. The patient will undergo a standard evaluation by a licensed respiratory therapist employed by Mount Sinai Hospital to develop the HBPR prescription. The evaluation will have two components, assessment of aerobic capacity using the 6-minute walk test (6MWT), and an assessment of muscular strength using elastic resistance bands. Target exercise intensity for HBPR will be set at 60-80% of the maximum work rate achieved during the 6MWT, a conservative goal intended to achieve benefit while minimizing risk of fatigue and shortness of breath. The therapist will select an appropriate band for home use for strength training exercises. During the evaluation, the respiratory therapist will monitor the patient's oxygen saturation, blood pressure, heart rate, and respiratory rate.

During the home visit that follows, the CHW will provide a timer, a pedometer to measure steps, an elastic resistance band, and an exercise diary. They may also provide the patient with an ergo cycle to enable them to conduct the aerobic exercises sitting down if walking is too burdensome or the patient is considered to be at high fall risk. The CHW and patient will consider the space available for exercise, such as a hallway, common space in the building (e.g., lobby, gathering room, etc.), outdoors during favorable weather, and local facilities like senior centers or churches. Once the area for exercise is selected, the CHW will demonstrate the walking and resistance training routines and observe the patient perform them on his/her own. The two will set a schedule for exercising and post the schedule and instructions prominently in the home.

Resistance training will consist of a simple routine of upper extremity extension and abduction movements with the elastic band. Each movement will be performed in 3 sets of 10 repetitions (15 minutes). The walking routine will last 20-40 minutes and the patient's pace will be guided by an audible click from the timer that is set by the CHW. The patient will be asked to perform the complete exercise routine 6 days a week. The CHW will directly supervise the patient multiple times over the 6-month intervention period. She will call periodically to support the patient when she is unable to visit.

The respiratory therapist will oversee the HBPR work of the CHW. This will include reviewing all cases in person or by phone every 7-14 days. Patients will be asked to reduce the intensity of exercise or rest for 5-10 minutes if they develop an uncomfortable level of shortness of breath or fatigue, and to stop exercising if they have symptoms that cause distress or discomfort and do not resolve after rest. Low literacy education methods will be used to ensure their understanding and retention of these instructions. The CHW will maintain communication with the therapist by HIPAA compliant secure email and telephone to report patient performance, trouble shoot problems, and to receive continuing education.

Step 7: Follow-up and Maintenance. The CHW will recommend that in-person meetings occur 1, 4, 8, and 12 weeks after intake and telephone follow-ups weekly through week 8 and monthly thereafter until month 6 when the intervention ends. Calls may be made more often to cognitively impaired patients to enhance information retention. Importantly, the patient and CHW will have the flexibility to tailor the number and frequency of encounters as they see fit. During follow up the CHW will assess patients' progress with SMB, their goals, and their symptoms.

Step 8: Graduation. SaMBA-COPD patients will receive a certificate upon program completion.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years
* Chart-document severe or very severe COPD (FEV1<50% predicted) or COPD-related ED/hospitalization ≥ 1 visit within the past 12 months
* Prescribed any daily medication for COPD, English or Spanish speaking, Smoking history ≥ 10 pack-years

Exclusion Criteria:

* Diagnosis in the clinical record of dementia, because the study focuses on patients with capacity to independently perform self-management tasks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected during the trial will not be shared.

REFERENCES:
- [Derived] Federman AD, Barry M, Moas E, Davenport C, McGeough C, Tejeda M, Rivera L, Gutierrez S, Mejias H, Belton D, Mathew C, Lindenauer PK, McDermott D, O'Conor R, Wolf MS, Wisnivesky JP. Protocol for a feasibility randomized trial of self-management support for people with chronic obstructive pulmonary disease using lay health coaches. Contemp Clin Trials. 2021 Nov;110:106570. doi: 10.1016/j.cct.2021.106570. Epub 2021 Sep 21. PMID 34560265
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Site for Phase 1: Icahn School of Medicine at Mount Sinai & Northwestern University, Phase 2 Site: Icahn School of Medicine at Mount Sinai
Period: Overall Study
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Started | 30 | 29
Completed | 28 | 24
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.7) | 64.0 (8.4) | 64.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 2 | 3 | 5
  Black, non-Hispanic | 17 | 11 | 28
  Hispanic | 11 | 15 | 26
Education [Count of Participants; unit: Participants]
  <High school | 10 | 8 | 18
  High school graduate | 7 | 9 | 16
  Some college | 9 | 10 | 19
  College graduate or higher degree | 3 | 2 | 5
  Missing information | 1 | 0 | 1
Number of participants with monthly household income ≤$3000 [Count of Participants; unit: Participants] | 26 | 24 | 50
Married/partnered [Count of Participants; unit: Participants] | 2 | 3 | 5
Number of participants with Medicaid insurance [Count of Participants; unit: Participants] | 19 | 19 | 38
Number of participants with marginal or inadequate Health Literacy [Count of Participants; unit: Participants] — Number of participants with marginal or inadequate health literacy. 3-item health literacy screen questions scored on a Likert scale from 0-4. Lower score indicates higher literacy. Variables were then dichotomized into Adequate health literacy (0,1) and Marginal/Inadequate health literacy (2,3,4)
  Participants | 16 | 14 | 30
Social Provisional Scale: The EPS-10 Items [Mean (Standard Deviation); unit: units on a scale] — The SPS-10 consists of 10 items, each item scored 4-point scale from 1 (strongly disagree) to 4 (strongly agree).
  The total SPS-10 score has a possible score range of 10-40, where a high score indicates high degree of social provisions..
  units on a scale | 32.7 (5.2) | 32.4 (4.0) | 32.6 (4.6)
Number of participants with poor-fair physical/mental general health on PROMIS Global Health (v 1.2) [Count of Participants; unit: Participants] — Number of participants with poor-fair physical/mental general health.
  PROMIS Global Health (v 1.2) - General health - categorized as Poor-Fair or Good-Very Good-Excellent.
  Participants | 9 | 7 | 16
Charlson Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — Charlson Comorbidity Index, age adjusted. Each condition is assigned a weight from 1 to 6, with full score from 0-37. Higher score indicates the higher the predicted mortality rate is.
  units on a scale | 6.0 (2.8) | 5.6 (2.6) | 5.8 (2.7)
Modified Activities of Daily Living (ADL) total score [Mean (Standard Deviation); unit: units on a scale] — ADL subscale 0-10, IADL subscale 0-14. Each item was re-coded as 0=independent, 1=needs some assistance, 2=cannot do without help. Total score 0-2. Higher score indicates more impairment.
  units on a scale | 0.7 (1.1) | 0.5 (1.2) | 0.6 (1.2)
Lawton -Brody Instrumental Activities of Daily Living Scale (IADL) total score [Mean (Standard Deviation); unit: units on a scale] — 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning).
  units on a scale | 2.3 (2.7) | 2.6 (2.5) | 2.5 (2.6)
Number of participants who scored between 11-21 on the HADS anxiety subscale [Count of Participants; unit: Participants] — Number of participants who scored between 11-21 on the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS).
  HADS is a 14-items scale with responses scored from 0-3, score range for anxiety subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more symptoms.
  Participants | 8 | 5 | 13
Number of participants who scored between 11-21 on the depression subscale of the HADS [Count of Participants; unit: Participants] — Number of participants who scored between 11-21 on the depression subscale of the HADS.
  HADS is a 14-items scale with responses scored from 0-3, score range for depression subscale is from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more symptoms.
  Participants | 3 | 4 | 7
Number of participants with for ≥mild impairment on the Trail Making Test B [Count of Participants; unit: Participants] — Number of participants with for ≥mild impairment
  The Trail Making Test is a performance based test of visual attention and task switching. Trails B requires the connection in sequence of 25 circles labeled by alternating numbers and letters (1-A-2-B-3-C). The score on the test is the time in seconds that it takes to complete. Higher time indicate poorer performance. The level of impairment is based on normative data adjusted t-scores (stratified by age and education). ≥ Mild impairment = ≥1 SD below mean.
  Participants | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: COPD Assessment Test (CAT)
Description: The COPD Assessment Test (CAT) is a validated measure designed to measure the impact of COPD on a person's life, and how this changes over time. Full range from 0-40, higher scores indicates a more severe impact of COPD on a patient's life.
Time Frame: Baseline and 6 months
Population: 6 month data provide for those who completed the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 30 | 29
score on a scale
  Baseline | 22.0 (8.6) | 21.9 (8.3)
  6 months: number analyzed (Participants) | 28 | 24
  6 months | 21.5 (9.6) | 22.7 (6.5)

2. Secondary Outcome: Number of Participants With Medication Adherence Report Scale (MARS) Score ≥4.5
Description: The MARS is a validated measure to assess COPD medication adherence. The MARS assess asthma beliefs about asthma medication adherence. The MARS is a 10-item instrument, full range from 0-10, higher score indicates higher likelihood of medication adherence.
  Adherence was defined as a score ≥4.5.
Time Frame: Baseline and 6 months
Population: Participants not included if not on controller medication or were not taking their prescribed controller medication/not filling doctor prescriptions and hence did not complete MARS.
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 29 | 27
Participants
  Baseline | 13 | 13
  6 months: number analyzed (Participants) | 28 | 22
  6 months | 14 | 10

3. Secondary Outcome: Exercise Tolerance - 6 Minute Walk Test
Description: The six minute walking test (6MWT), developed by the American Thoracic Society, is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes. Participants walked back and forth in the hallway with aim to walk as far as possible in 6 minutes. Participants were allowed to slow down, to stop, and to rest as necessary. They may stand and rest but resume walking as soon as they were able.
Time Frame: Baseline and 6 months
Population: Reasons for missed visits include 6 month phone interview instead of in person visit, participants not feeling well or wheelchair bound.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 26 | 25
meters
  Baseline | 244.3 (92.4) | 288.3 (101.2)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 266.9 (76.9) | 291.0 (68.8)

4. Secondary Outcome: Physical Activity Adult Questionnaire (PAAQ)
Description: The PAAQ captures behavior in the seven days before the visit. Questions pertain to total time spent doing moderate to vigorous-intensity physical activity (MVPA) in three domains: transportation, leisure time and other (includes work, home and volunteering), and how much time was dedicated to vigorous activity (compared with total MVPA). Respondents are asked to report activities that lasted at least 10 consecutive minutes.
  Once completed, a total amount of time spent doing MVPA in the last 7 days was calculated.
  Cut off in terms of the specific definition of physical activity in the Guidelines->accumulating at least 150 minutes of MVPA a week in bouts of at least 10 minutes is considered adequate.
Time Frame: Baseline and 6 months
Population: Missing data because there is branching logic in instrument, wherein, if the previous question asking whether an activity was done is answered "no", the following question will not be asked to the participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 20 | 21
minutes
  Baseline | 214 (190) | 231 (294)
  6 months: number analyzed (Participants) | 20 | 15
  6 months | 262 (271) | 234 (402)

5. Secondary Outcome: Number of Participants With Hospitalizations
Description: Number of participants with hospitalizations for COPD exacerbations or any respiratory issue in the prior 6 months.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 30 | 29
Participants
  Baseline | 15 | 14
  6 months | 10 | 12

6. Secondary Outcome: Number of Participants With ED Visits
Description: Number of participants with Emergency Dept (ED) for COPD exacerbations or any respiratory issue in the prior 6 months.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 30 | 29
Participants
  Baseline | 15 | 19
  6 months | 13 | 13

7. Secondary Outcome: Number of Participants With Controller Medication Adherence
Description: Medication adherence was also measured using electronic monitoring devices, the Doser CT (Meditrack, Hudson, MA) for metered dose inhalers and the Smartdisk (Nexus6, Franklin, OH) for dry powder inhalers. Patients used the devices over a 4-week period of observation. Adherence was defined as use of ≥80% of doses prescribed.
Time Frame: Baseline and 6 months
Population: Data for participants that have controller device data
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
Number analyzed (Participants) | 13 | 11
Participants
  Baseline: number analyzed (Participants) | 9 | 11
  Baseline | 3 | 3
  6 months: number analyzed (Participants) | 13 | 8
  6 months | 5 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Targeted Self-management Barrier Support | Guided COPD Education
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04533412/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT04533412/SAP_001.pdf
  • Informed Consent Form (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04533412/ICF_002.pdf